CLINICAL TRIAL: NCT02407314
Title: Impact of Ticagrelor and Aspirin Versus Clopidogrel and Aspirin in Patients With Claudication and Peripheral Arterial Disease (PAD): Thrombus Burden Assessed by Optical Coherence Tomography
Brief Title: Ticagrelor and Peripheral Arterial Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: AZ discontinued study
Sponsor: Arkansas Heart Hospital (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10020
Record Dates: First submitted 2015-03-18; First posted 2015-04-02 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Optical Coherence Tomography; Ticagrelor; Aspirin; Claudication; Clopidogrel
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Tomography, Optical Coherence; Aspirin; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin only (Sham Comparator): Clopidogrel 75 mg + aspirin 81 mg for the first month followed by aspirin 81 mg alone for months 2-6 months post percutaneous peripheral intervention (PPI) intervention assessed by optical coherence tomography (OCT) ankle brachial index (ABI) and six minute walk distance.
  Interventions: Procedure: Percutaneous Peripheral Intervention; Device: Optical Coherence Tomography; Other: Ankle Brachial Index; Other: Six minute walk distance; Drug: Aspirin
- Aspirin + Ticagrelor (Experimental): ticagrelor 90 mg bid + aspirin 81 mg for months 1-6 months post percutaneous peripheral intervention (PPI) intervention assessed by optical coherence tomography (OCT)ankle brachial index (ABI) and six minute walk distance.
  Interventions: Procedure: Percutaneous Peripheral Intervention; Device: Optical Coherence Tomography; Other: Ankle Brachial Index; Other: Six minute walk distance; Drug: Aspirin + Ticagrelor

INTERVENTIONS:
Procedure: Percutaneous Peripheral Intervention — Percutaneous peripheral intervention is a common procedure performed by cardiologists to revascularize peripheral arterial lesions in patients (stent placement). This procedure is considered standard of care and is not experimental.
Device: Optical Coherence Tomography — This is an established medical imaging technique that uses light to capture micrometer-resolution, three-dimensional images from within optical scattering media. The device used is a cardiac catheter with OCT sensors on the tip of it. It will be used to assess the artery vessels after Percutaneous Peripheral Intervention.
Other: Ankle Brachial Index — This a clinical assessment and consists of the calculation of the ratio of the blood pressure in the lower legs to the blood pressure in the arms. The ABI is calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressures in the arm.
Other: Six minute walk distance — Assessment of the walking distance in 6 minutes.
Drug: Aspirin — Aspirin, also known as acetylsalicylic acid [ASA], is a salicylate drug, often used as an analgesic to relieve minor aches and pains, as an antipyretic to reduce fever, and as an anti-inflammatory medication. Aspirin also has an antiplatelet effect by inhibiting the production of thromboxane, which under normal circumstances binds platelet molecules together to create a patch over damaged walls of blood vessels.
  Other Names: Acetylsalicylic acid [ASA]
  Arms: Aspirin only
Drug: Aspirin + Ticagrelor — This is a combination of drugs (Aspirin + Ticagrelor). Ticagrelor is a platelet aggregation inhibitor due to its properties as an antagonist of the P2Y12 receptor. Ticagrelor is a nucleoside analogue: the cyclopentane ring is similar to the sugar ribose, and the nitrogen rich aromatic ring system resembles the nucleobase purine, giving the molecule an overall similarity to adenosine.
  Other Names: acetylsalicylic acid [ASA] + Brillinta
  Arms: Aspirin + Ticagrelor

SUMMARY:
This is an interventional study assessing the effectiveness of Ticagrelor on the reduction of thrombus burden using optical coherence tomography in patients undergoing peripheral artery stenting.

DETAILED DESCRIPTION:
Prospective, randomized study, comparing ticagrelor + aspirin vs. aspirin monotherapy following the 4-week post-procedural combination of Ticagrelor or Plavix with low dose aspirin. The investigators will enroll a minimum of 40 patients. Patients will be enrolled if they have either claudication and/or critical limb ischemia, and angiographically identified superficial femoral artery (SFA) disease requiring intervention, with either total occlusion or a significant SFA stenosis with the presence of Optical Coherence Tomography (OCT) defined clot following stent placement.

Participants will be evaluated at baseline, 1 month, 4 months, 6 and 7 months following SFA intervention. At baseline demographic data will be collected, and anthropomorphic and physiological variables (body mass index, waist circumference, blood pressure). Baseline and 6-month ankle brachial index (ABI) will be performed. A 6-min walk test will be performed at baseline and 6-month follow-up. At 6 month time point patients in both treatment groups will return for a peripheral angiogram and repeat OCT imaging of the SFA segments of interest. Subject will have a final follow up clinic visit at 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower extremity claudication and PAD due to significant SFA stenosis (>60%) or total occlusions (Rutherford 2-6) that affects the quality of life despite medical therapy.
* The presence of OCT identified clot in the Superficial Femoral Artery (SFA) following stent placement.
* Evidence of significant SFA disease involving the most symptomatic limb established by noninvasive vascular testing (ankle-brachial index [ABI] <0.9, toe brachial Index [TBI] of <0.6. If ABI>1.4, SFA systolic acceleration time >140 milliseconds); computed tomographic angiography, or magnetic resonance angiography confirming at least a 60% stenosis of the SFA.
* At least one non-treated Below The Knee (BTK) vessel patent
* Male and female outpatients 18 years of age.
* The only following devices may be used for the revascularization procedures: conventional balloons and bare metal stents (block randomization).
* Subject has been advised of the beneficial effects of smoking cessation and regular exercise but must not be in the process of changing their smoking status at the time of screening. Patients may resume or increase exercising as an effect of post procedurally improved lower limb perfusion.
* Peak Walking Time (PWT) limited only by claudication.
* Willingness to participate, documented by written informed consent.

Exclusion Criteria:

* Patients requiring dual anti-platelet drug treatment before start of study
* Planned amputation
* Use of atherectomy devices
* Hypersensitivity to acetylsalicylic acid, or ticagrelor. For ticagrelor, hypersensitivity reactions in the past include angioedema
* Patients with known bleeding disorders
* Patients with known active pathological bleeding
* Patients needing chronic oral anticoagulant maintenance therapy
* Patients with a history of intracranial hemorrhage at any time, GI bleed in the past 6 months, or major surgery within the past 30 days
* Ischemic stroke during the past 3 months
* Patients considered to be at risk of bradycardic events unless treated with a permanent pacemaker
* Target is a restenotic lesion or in-stent restenosis
* Any scheduled revascularization procedure requiring dual-anti-platelet therapy for more than one month
* Severe hypertension that may put the patient at risk, systolic greater than or equal to 180 and/or diastolic greater than or equal to 100
* Severe liver disease
* History of congestive heart failure with an Left Ventricular Ejection Fraction (LVEF) of less than 30%
* Concern for inability of the patient to comply with study procedures and/or follow up (eg, alcohol or drug abuse)
* Infra-popliteal disease involving the last remaining vessel (single run-off)
* Prior lower extremity revascularization within the past 30 days prior to enrollment
* Atherectomy of PAD
* EXCIPIENTS to ticagrelor hypersensitivity
* Known pregnancy, breast-feeding, or intend to become pregnant during the study period (all female patients 55 years and younger, without past history of hysterectomy must have a pregnancy test prior to peripheral intervention at baseline and at 6 months)
* Creatinine clearance < 30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Change in the Intraluminal clot volume (in mm3) | At baseline and at 6 months
  Intraluminal clot volume will be assessed by Optical Coherence Tomography using a Core Lab.
Change in the Intraluminal clot length (mm) | At baseline and at 6 months
  Intraluminal clotlength will be assessed by Optical Coherence Tomography using a Core Lab.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Cilingiroglu, MD, Principal Investigator — Arkansas Heart Hospital; Massoud Leesar, MD, Principal Investigator — University of Alabama at Birmingham; Hinan Ahmed, MD, Principal Investigator — University Of Texas Health Science Center in San Antonio; Marc D Feldman, MD, Principal Investigator — University Of Texas Health Science Center in San Antonio; Gerardo Rodriguez, MD PhD, Study Director — Arkansas Heart Hospital
Locations (1):
- Arkansas Heart Hospital, Little Rock, Arkansas, United States